CLINICAL TRIAL: NCT03848013
Title: Reatment of Melasma Using Q-switched Nd: YAG Laser and Fractional CO2 Laser Separately and in Combination
Brief Title: Treatment of Melasma Using Q-switched Nd: YAG Laser and Fractional CO2 Laser Separately and in Combination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rana F Hilal, MD, Lecturer of dermatology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoU
Record Dates: First submitted 2018-12-12; First posted 2019-02-20 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Treatment of cases of melasma using Q switched Nd YAG laser and Fractional CO2 laser separately and in combination
  Interventions: Device: Q switched Nd YAG laser; Device: Fractional CO2 laser
- Follow -up period (No Intervention): follow up of the treated cases for 2 months

INTERVENTIONS:
Device: Q switched Nd YAG laser — Laser device emitting Q switched Nd YAG aiming for skin toning
  Arms: Treatment
Device: Fractional CO2 laser — Laser device emitting fractionated ablative laser aiming for skin resurfacing
  Arms: Treatment

SUMMARY:
* All participants will be divided into 2 groups : Group A & Group B.
* Group A will be subjected to 3 consecutive sessions of Q-switched 1,064 nm Nd: YAG laser to one side of the face & fractional co2 laser to the other side of the face with one month interval between sessions.
* Group B will be subjected also to 3 consecutive sessions of Q-switched 1,064 nm Nd: YAG laser to one side of the face & an additional fractional co2 laser to the other side of the face using the above mentioned parameters with one month interval between sessions.
* Response to treatment will be assessed using the Melanin Index (MI) score, Melasma Area and Severity Index (MASI) score, spectrophotometer ( Derma catch, colorix, Neuchatel, Switzerland ) and a subjective self-assessment method.

ELIGIBILITY:
Inclusion Criteria:

* melasma patients above 18 years

Exclusion Criteria:

* Pregnancy.
* Usage of chemical peeling 1 month prior to the study.
* Isotretinoin intake 6 months prior to the study.
* Any laser procedure related to melasma lesions 1 month prior to the study.
* Active herpetic lesions.
* Any concurrent active skin disease within the treated area.
* Photosensitive skin conditions such as systemic lupus erythematous.
* History of delayed wound healing.
* Keloid formation.
* Bleeding diathesis.
* Medical conditions such as diabetes mellitus & autoimmune diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Modified Melasma Area and Severity index change. | 6 months to 1 year
  Evaluate the efficacy of Q-switched 1,064nm Nd: YAG & fractional Co2 laser in the treatment of melasma by comparing the results through measuring modified MASI score before treatment and after treatment and follow-p period.
Melanin index change. | 6 months to 1 year
  Evaluate the efficacy of Q-switched 1,064nm Nd: YAG & fractional Co2 laser in the treatment of melasma by comparing the results by taking spectrophotometer readings (melanin index) before treatment and after treatment and follow-p period.
percentage of clinical improvement | 6 months to 1 year
  Evaluate the efficacy of Q-switched 1,064nm Nd: YAG & fractional Co2 laser in the treatment of melasma by comparing the results of masked dermatologists' observation of clinical photographs before treatment and after treatment and follow-p period.
patient satisfaction rate | 6 months to 1 year
  Evaluate the efficacy of Q-switched 1,064nm Nd: YAG & fractional Co2 laser in the treatment of melasma by comparing patient satisfaction before treatment and after treatment and follow-p period.

SECONDARY OUTCOMES:
Modified Melasma Area and Severity Index change. | 6 months to 1 year
  Evaluate the role of additional fractional co2 laser to the previously Q switched Nd: YAG treated melasma patients by measuring changes in modified MASI score before treatment and after treatment and follow-p period.
Melanin index change. | 6 months to 1 year
  Evaluate the role of additional fractional co2 laser to the previously Q switched Nd: YAG treated melasma patients by taking spectrophotometer readings (melanin index) before treatment and after treatment and follow-p period.
percentage of clinical improvement | 6 months to 1 year
  Evaluate the role of additional fractional co2 laser to the previously Q switched Nd: YAG treated melasma patients by comparing the results of masked dermatologists' observation of clinical photographs before treatment and after treatment and follow-p period.
patient satisfaction rate | 6 months to 1 year
  Evaluate the role of additional fractional co2 laser to the previously Q switched Nd: YAG treated melasma patients by comparing patient satisfaction before treatment and after treatment and follow-p period.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Kasr Al Ainy Hospital Dermatology department, Cairo, El Manial, Egypt